CLINICAL TRIAL: NCT06001801
Title: Leveraging Peer Support and Vouchers for Healthy Food to Increase Engagement in Diabetes Prevention Behaviors Among Low-income Adults With Prediabetes: the INSPIRing Action to Prevent Diabetes (INSPIRA) Intervention
Brief Title: The Inspiring Action to Prevent Diabetes Intervention
Acronym: INSPIRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Mary Ellen Michele Heisler, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00227197
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: PreDiabetes
Keywords: Diabetes Prevention Program; Behaviors; Weight loss; Healthy lifestyle changes; Peer Partner
MeSH Terms: conditions — Prediabetic State; Behavior; Weight Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Program (DPP) (usual care) (Active Comparator)
  Interventions: Behavioral: Diabetes Prevention Program
- DPP plus the INSPIRA intervention (Experimental): This arm will include the DPP plus additional interventions.
  Interventions: Behavioral: Diabetes Prevention Program; Behavioral: INSPIRA

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — The DPP group is led by the Community Health and Social Services Center (CHASS) community health workers (CHWs). For this study, the workers will deliver 16 weekly sessions (core phase) followed by two monthly sessions (maintenance phase). Each session lasts one hour plus the time required to weigh each participant and review food and activity logs.
  This program will help participants make healthy lifestyle changes. Examples are improvements in eating and physical activity. The goal is that participants lose some weight and eat healthier food.
  Sessions will be offered in-person in a room with video capacity to allow attendance of participants that cannot attend in person. For those participating virtually, the CHWs will briefly review with them what participants logged.
  Participation in this project should last approximately 6-months.
Behavioral: INSPIRA — This intervention will include the DPP plus additional interventions. The additional interventions include: participants to stay for an extra 30 minutes following the regular DPP sessions. In these INSPIRA sessions, participants will be trained in providing mutual peer support, be matched with a peer partner and asked to talk at least once a week, receive vouchers or gift cards, discuss participants action plans with the peer partner, and share challenges, successes, and tips from the CHW and others in the session.
  CHWs will provide brief trainings on autonomy-supportive peer support approaches over the first three weeks of sessions.
  Participation in this project should last approximately 6-months.
  Arms: DPP plus the INSPIRA intervention

SUMMARY:
This research is studying how to help increase uptake of and engagement in formal Diabetes Prevention Programs to improve healthy behaviors among adults with pre diabetes to reduce risk of getting diabetes.

This project will compare the Diabetes Prevention Program (DPP) to participating in the DPP program plus two extra pieces (INSPIRA). The 2 additional pieces in the DPP plus program includes getting matched with someone else in the program to provide each other support along with a chance to earn healthy food vouchers.

Eligible participants will be randomized to one of the two groups and be asked to participate for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking
* Body Mass Index (BMI) > 24.9 kilograms/meters squared (kg/m2)
* The most recent A1c test, completed in 60 days or fewer prior to enrollment, is 5.7%-6.4%

Exclusion Criteria:

* Diagnosed with schizophrenia
* Active alcohol or other drug abuse
* Are pregnant or planning pregnancy in next 6 months
* Will not be in local area in six months
* Will not be able to attend sessions, in-person or remotely, for three more weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of group sessions attended by participants | 6 months
  This count will be out of 16 possible weekly group sessions.

SECONDARY OUTCOMES:
Change in weight | baseline, 6 months
  Weight will be measured in pounds to the nearest tenth.
Change in hemoglobin A1c | baseline, 6 months
Change in waist circumference | baseline, 6 months
  This will be measured in centimeters.
Change in reported diet quality | baseline, 6 months
  measured by comparing baseline and six month survey responses

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen M Heisler, MD, Principal Investigator — University of Michigan
Locations (1):
- Community Health and Social Services Center, Incorporated, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT06001801/ICF_000.pdf